CLINICAL TRIAL: NCT03472820
Title: The Effects of Diet and Lifestyle on Quality of Life and Methylation-related Biomarkers in Vivo.
Brief Title: Methylation Diet and Lifestyle Study
Acronym: MDL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Dr. Kara Fitzgerald, ND (Unknown); Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RB100217
Record Dates: First submitted 2018-02-22; First posted 2018-03-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Lifestyle; Diet; Healthy
Keywords: Diet; Lifestyle; DNA methylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention will be diet, lifestyle, exercise and stress management recommendations combined with taking two different supplements twice daily, in divided doses.
  Interventions: Other: Diet Recommendations; Other: Lifestyle Recommendations; Other: Exercise Recommendations; Other: Stress Management Recommendations; Other: PhytoGanix (tropical fruit flavor); Other: UltraFlora Intensive Care
- Control Group (No Intervention): The control group will undergo the same testing measures as the intervention group, but will not have access to the education information or be instructed to change diet or lifestyle factors. They will have access to the information after the study is complete.

INTERVENTIONS:
Other: Diet Recommendations — Specific dietary guidelines will be outlined for participants.
  Arms: Intervention Group
Other: Lifestyle Recommendations — Participants are encouraged to average a minimum of 7 hours of sleep per night.
  Arms: Intervention Group
Other: Exercise Recommendations — Participants will be encouraged to exercise a minimum of 30 minutes at least 5 days per week at an intensity of 60-80% of maximum perceived exertion.
  Arms: Intervention Group
Other: Stress Management Recommendations — Participants will utilize the Cleveland Clinic's Stress Free Now application to engage in a variety of guided stress reduction techniques, including meditation and mindful breathing. Recommended frequency is twice daily, preferably morning and evening.
  Arms: Intervention Group
Other: PhytoGanix (tropical fruit flavor) — Organic Superfruits & Greens Powder Drink Mix is a food-based phytonutrient blend. Participants will take 2 servings daily in divided doses.
  Arms: Intervention Group
Other: UltraFlora Intensive Care — Probiotic; Participants will take 2 capsules of UltraFlora Intensive Care probiotic daily in divided doses.
  Arms: Intervention Group

SUMMARY:
The maintenance of health and the progression of disease are associated with an individual's genetic make-up and environmental factors, including lifestyle choices (such as diet, exercise, behaviors, stressors, sleep, tobacco and alcohol use), environmental exposures and socioeconomic determinants. Environmental factors have been shown to influence, sometimes rapidly, epigenetic processes thereby influencing genetic expression. Regulation of the human genome by the epigenome is now regarded as a cornerstone, heritable, physiologic process, playing a key role in phenotypic expression of health and disease.

DNA methylation is a well-researched, primary epigenetic process. Aberrant DNA methylation resulting in hyper- or hypomethylated regions of the genome, generally results in inhibition or expression of certain genes and has been associated with the pathogenesis of numerous conditions, ranging from inflammation and accelerated aging, to cancer, autoimmunity, diabetes, heart disease, dementia, allergic disease, posttraumatic stress disease and others. Likewise, certain healthy diet and lifestyle habits have been demonstrated to favorably influence DNA methylation patterns.

Understanding that environmental factors can potently and sometimes rapidly, favorably or negatively influence epigenetic expression, a short-term diet and lifestyle intervention may significantly augment DNA methylation expression.

The purpose of this study is to evaluate a 9-week diet and lifestyle intervention on patient-reported quality of life, symptoms, and DNA and biochemical methylation-related biomarkers in healthy males ages 50-72.

ELIGIBILITY:
Inclusion Criteria:

* • Males, ages 50-72

  * Willing to adhere to 9 weeks of a dietary and lifestyle program including specific nutrition and exercise guidelines
  * Willing to avoid any over-the-counter medications, supplements or herbal products for the length of the study, except short-term use (<1 week) use at least 1 week before scheduled study visits
  * Willing to have blood drawn three times and abstain from food or beverage intake for 10-12 hours before blood draws
  * Willing to provide saliva samples
  * Willing to track food intake, sleep, stress management techniques, and exercise daily
  * Willing to drink a nutrient-enriched beverage and take a encapsulated probiotic daily
  * Willing and able to use electronic devices and connect to the internet
  * Able to speak, read and understand English

Exclusion Criteria:

* • Currently taking any of the following prescription medications

  * Proton pump inhibitors: omeprazole (Prilosec, Prilosec OTC); aspirin and omeprazole (Yosprala); lansoprazole (Prevacid, Prevacid IV, Prevacid 24-Hour); ;dexlansoprazole (Dexilent, Dexilent Solutab); rabeprazole (Aciphex, Aciphex Sprinkle); pantoprazole (Protonix)
  * H2-blockers: nizatidine (Axid, Axid AR, Axid Pulvules); famotidine (Pepcid, Pepcid AC); cimetidine (Tagamet, Tagamet HB); ranitidine (Zantac)
  * These classes of medications are excluded due to direct (due to nutrient requirements for metabolism) and indirect (through impaired digestion and assimilation of nutrients).

    * Use of nutrition supplements or herbal products not prescribed by a licensed healthcare provider for a medical condition
    * Currently following a prescribed dietary/lifestyle program or initiate within the 30 days prior to baseline
    * Initiation of or changes to an exercise regimen within 30 days prior to baseline
    * Use of nicotine, marijuana or cannabinoids (including CBD products) or recreational drugs/substances (such as but not limited to cocaine, phencyclidine [PCP], and methamphetamine) current/within the last 30 days or use during the study
    * Have a diagnosis of cardiovascular disease, kidney disease, liver disease, diabetes, autoimmune disease, high blood pressure, or cancer (does not include basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix).
    * Have a diagnosis of an immunodeficiency condition, such as Human Immunodeficiency Virus (HIV) infection or Acquired Immune Deficiency Syndrome (AIDS)
    * Have a diagnosis of neurodegenerative conditions such as, amyotrophic lateral sclerosis (ALS), Parkinson's disease, Multiple Sclerosis, or Alzheimer's disease.
    * Excessive alcohol consumption (more than 4 drinks per day or 14 per week on average)
    * Known sensitivity, intolerance or allergy to ingredients in the study supplements or in the recommended dietary therapy
    * Currently receiving intravenous nutrient therapy
    * Currently participating in another interventional research study or participated in another interventional study within the last 3 weeks prior to baseline

Ages: 50 Years to 72 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 44 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) | 8 weeks
  PROMIS-29 will measure health-related quality of life and is a validated, 29 question survey divided into seven sub-domains of function including physical functioning, social function, pain interference, pain intensity, sleep, depression, and anxiety.

SECONDARY OUTCOMES:
Measure Yourself Medical Outcome Profile (MYMOP) | 8 weeks
  MYMOP will measure change(s) in patient-reported symptoms and is a patient-centered outcome measure that allows for the participant to self-select their top health concern(s) or symptom(s) they are dealing with in their own words. The participant can also choose an activity that is limited by that health concern.
National University of Natural Medicine Multi-system Symptom/Adverse Event Questionnaire | 8 weeks
  The NUNM Multi-system Symptom/Adverse Event Questionnaire measures change(s) in patient-reported symptoms and is a standardized ninety-one point monitoring form that requires asking questions pertaining to the following organ systems: eyes/ears/nose/throat, gastrointestinal, neurological/ musculoskeletal, psychological/general, cardiopulmonary, skin, genitourinary and whole body systems.

OTHER OUTCOMES:
Infinium Methylation EPIC Index by Illumina | 8 weeks
  Infinium Methylation EPIC Index by Illumina measures the methylation status of CpG sites. Epigenetic profile that assesses methylation on over 850,000 CpG DNA sites. A saliva sample will collect approximately 2 mL (~1 teaspoon) into a cryovial.
Methylation Profile by Doctor's Data | 8 weeks
  Methylation Profile by Doctor's Data measures the changes in the methylation related biomarkers and is a functional assessment of the phenotypic expression of common single nucleotide polymorphisms (SNPs) and provides a "methylation index," a ratio of S-Adenosylmethionine (SAM) to S-Adenosylhomocysteine (SAH).
Folate Vitamer Panel by Doctor's Data | 8 weeks
  Folate Vitamer Panel by Doctor's Data measures the changes in the methylation related biomarkers and measures folate congeners affecting enzyme function in methylation pathways including unmodified Folic Acid (UMFA), 5-Methyltetrahydrofolate (5-MTHF), tetrahydrofolate (THF), folinic Acid (5-CHO-THF).
Medical Symptom Questionnaire (MSQ) | 8 weeks
  The MSQ measures change(s) in patient-reported symptoms and is a 71-question measure that measures various health areas including: Digestive tract, Eyes, Energy/Activity, Emotions, Head, Heart, Joint/Muscles, Lungs, Mind, Mouth/Throat, Nose, Skin, Weight, and Other.
DNA Methylation Pathway Profile by Doctor's Data | 8 weeks
  DNA Methylation Pathway Profile is a measurement of potential confounders and assesses changes to single nucleotide polymorphisms (SNPs) - DNA genotype which may affect enzymatic function which include, methionine metabolism, detoxification, hormones, and vitamin D. This is a blood spot test and requires collection of 5 drops of blood after a finger stick.

CONTACTS AND LOCATIONS:
Locations (1):
- NUNM Helfgott Research Institute, Portland, Oregon, United States

DOCUMENTS (1):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT03472820/Prot_000.pdf